CLINICAL TRIAL: NCT06681285
Title: The Efficacy and Safety of Cadonilimab Combined With Anlotinib Followed by Radiotherapy in the Second and Later-line Treatment of Recurrent or Metastatic Esophageal Squamous Cell Carcinoma (CAR-RMEC):A Single-arm, Multicenter, Phase II Clinical Trial
Brief Title: Cadonilimab Combined With Anlotinib Followed by Radiotherapy in Recurrent or Metastatic Esophageal Squamous Cell Carcinoma (CAR-RMEC)
Acronym: CAR-RMEC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024207
Record Dates: First submitted 2024-11-01; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Carcinoma
Keywords: Cadonilimab; Anlotinib; Radiotherapy; Esophageal carcinoma
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab Combined With Anlotinib Followed by Radiotherapy in the Second and Later-line Treatment (Experimental): Cadonilimab Combined With Anlotinib Followed by Radiotherapy in the Second and Later-line Treatment of Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
  Interventions: Drug: Cadonilimab ;Anlotinib

INTERVENTIONS:
Drug: Cadonilimab ;Anlotinib — Cadonilimab Combined With Anlotinib Followed by Radiotherapy in the Second and Later-line Treatment of Recurrent or Metastatic Esophageal Squamous Cell Carcinoma

SUMMARY:
GLOBOCAN 2020 reported that the global incidence of esophageal cancer climbed to 604,100, accounting for 3.1% of all tumor sites and ranking 7th out of 36 cancers. In addition, about 544,076 new esophageal cancer deaths, which accounted for 5.5% of all study centers and ranked 6th among 36 cancers. Esophageal squamous cell carcinoma (ESCC) is the most common pathological type of esophageal cancer in China, and accounts for about 90% of cases. Immunotherapy has become the main treatment for second-line and later esophageal cancer patients, but because of the single target, limited mediated signaling pathway, and high drug resistance rate, single-target blocking has limited efficacy. Cadonilimab is a novel humanized bispecific antibody targeted by programmed death receptor 1（PD-1）/cytotoxic T-lymphocyte antigen 4 (CTLA-4)，which can simultaneously block the two immune checkpoint pathways of PD-1 and CTLA-4, indirectly "liberating" immune cells, and improving immune efficacy. Anlotinib inhibits tumor angiogenesis by fully acting on the VEGFR/PDGFR/FGFR pathway, while remodeling tumor microenvironment, increasing T cell activity and infiltration, and synergizing immunotherapy. In addition, the control of local tumors or oligometastases by radiotherapy combined with systemic therapy such as immunotherapy has become an important research direction for metastatic esophageal cancer. This study will explore the efficacy and safety of cadonilimab combined with anlotinib sequential radiotherapy for the treatment of recurrent or metastatic esophageal squamous cell carcinoma (ESCC) at second or later line.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up;
2. Patients with recurrent/metastatic esophageal squamous cell carcinoma were confirmed by pathology or cytology.
3. Age≥18 years old, male or female;
4. Eastern Cooperative Oncology Group（ECOG） score 0-2 points;
5. Patients who have not received systematic treatment for recurrent/metastatic esophageal squamous cell carcinoma or have received systematic treatment failure for recurrent/metastatic esophageal squamous cell carcinoma;
6. According to the solid tumor efficacy evaluation criteria (RECIST version 1.1), there is at least one radiographically measurable lesion;
7. Expected survival time ≥3 months;
8. There is sufficient organ and bone marrow function, as follows:

   1. Hemoglobin (Hb) ≥ 90g/L;
   2. Neutrophil count (ANC) ≥ 1.5 × 109/L;
   3. Platelet count (PLT) ≥ 100 × 109/L;
   4. Serum albumin (ALB) ≥ 30g/L;
   5. Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 ULN; If there is liver metastasis, ALT and AST should be ≤ 5ULN;
   6. Total bilirubin (TBIL) ≤ 1.5ULN;
   7. Serum creatinine (Cr) ≤ 1.5ULN or creatinine clearance rate (CCr) ≥ 60ml/min;
   8. International normalized ratio (INR) ≤ 1.5, activated partial thromboplastin time (APTT) ≤ 1.5 times ULN;
   9. Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
   10. The myocardial enzyme spectrum is within the normal range (simple laboratory abnormalities that are deemed clinically insignificant by the researchers are also allowed to be included);
9. Echocardiographic evaluation: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%);
10. Women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, birth control pills, or condoms) during the study period and within 6 months after the end of the study; Within 7 days prior to enrollment in the study, the serum or urine pregnancy test must be negative and the patient must be non lactating; Men should agree to use contraception during the study period and for 6 months after the end of the study period for patients

Exclusion Criteria:

1. Patients with uncontrolled or symptomatic active central nervous system (CNS) metastases (patients with CNS metastases who have been adequately treated, are clinically stable for at least 2 weeks, and have stopped corticosteroids 1 week prior to enrollment can be enrolled, and patients with asymptomatic BMS who do not require treatment can be enrolled);
2. There is pleural or peritoneal effusion or pericardial effusion that cannot be controlled after effective treatment;
3. Patients with serious concurrent diseases, such as heart failure, high-risk uncontrolled arrhythmias, severe myocardial infarction, refractory hypertension, renal failure (CKD-stage 4 and above), thyroid insufficiency, mental illness, diabetes, severe chronic diarrhea (more than 7 defecation times per day), etc., and who are deemed unsuitable for participation in this clinical study by the researchers;
4. The presence of any active, known or suspected autoimmune disease. Admitted subjects who are in a stable state and do not require systemic immunosuppressive therapy;
5. Any other malignancies developed during the first 3 years of study, except locally treatable and cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, breast ductal carcinoma in situ, and papillary thyroid cancer
6. human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as HBV-DNA≥1000 copies /ml; Hepatitis C, defined as HCV-RNA above the lower detection limit of analytical methods) or co-infection with hepatitis B and hepatitis C;
7. Imaging during the screening period showed that the tumor surrounded or invaded important blood vessels or organs (such as the heart and pericardium, trachea, aorta, superior vena cava, etc.) or had obvious necrosis and voids, and the researchers determined that entering the study would cause bleeding risk; Subjects at risk for esophagotracheal or esophagopleural fistula；
8. Past or current non infectious pneumonia/interstitial lung disease (including radiation pneumonitis) requiring systemic corticosteroid therapy;
9. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
10. Individuals who are allergic to the drugs or their components used in this program;
11. Any of the following situations occurred during previous PD-1 inhibitor treatment:

    1. Previous occurrence of grade 3 or higher immune-related adverse events(irAE )(excluding endocrine system related irAE) resulting from PD-1 inhibitor therapy, irAE resulting in permanent discontinuation of therapy, grade 2 immune-related cardiotoxicity, or neurological or ocular irAE of any grade.
    2. Prior to screening in this study, all adverse events treated with prephase PD-1 inhibitors had not been fully resolved or had not been resolved to grade 1. Subjects with grade 2 or greater endocrine adverse events were admitted if their condition was stable and asymptomatic with appropriate alternative therapy.
    3. Prior adverse events requiring immunosuppressant therapy other than glucocorticoids, or recurrent adverse events during prior immunotherapy requiring systemic glucocorticoid therapy;
12. Pregnant or lactating women;
13. with a history of psychiatric drug abuse and can not quit or patients with mental disorders;
14. The researcher thinks that it is not appropriate to participate in this researcher; 15, unwilling to participate in the study or unable to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of progression-free survival (PFS) in Second and Later-line Treatment of Recurrent or Metastatic Esophageal Squamous Cell Carcinoma patients receiving Cadonilimab Combined With Anlotinib Followed by Radiotherapy | 2 years
  PFS is defined as the time from the start of enrollment until tumor progression or death from any cause.

SECONDARY OUTCOMES:
Assessment of objective remission rate (ORR) in the Second and Later-line Treatment of Recurrent or Metastatic Esophageal Squamous Cell Carcinoma patients receiving Cadonilimab Combined With Anlotinib Followed by Radiotherapy | 2 years
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Objective remission rate (ORR): defined as the proportion of subjects whose tumor volume shrinks to a pre-specified value and can be maintained for the minimum time frame required, incorporating cases in complete remission (CR) and partial remission (PR).
Assessment of disease control rate (DCR) in the Second and Later-line Treatment of Recurrent or Metastatic Esophageal Squamous Cell Carcinoma patients receiving Cadonilimab Combined With Anlotinib Followed by Radiotherapy | 2 years
  Disease control rate (DCR): the proportion of patients whose tumors shrank or were stable and remained so for a certain period of time, including complete remission (CR), partial remission (PR) and stable disease (SD)
Assessment of overall survival (OS) in the Second and Later-line Treatment of Recurrent or Metastatic Esophageal Squamous Cell Carcinoma patients receiving Cadonilimab Combined With Anlotinib Followed by Radiotherapy | 2 years
  OS is defined as the time from the start of enrollment to death from any cause.

OTHER OUTCOMES:
Assessment of the incidence of treatment-related adverse evants in the Second and Later-line Treatment of Recurrent or Metastatic Esophageal Squamous Cell Carcinoma patients receiving Cadonilimab Combined With Anlotinib Followed by Radiotherapy | 2 years
  Adverse events are observed during the course of the study and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE V5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China